CLINICAL TRIAL: NCT02454972
Title: A Multicenter Phase II Clinical Trial of Lurbinectedin (PM01183) in Selected Advanced Solid Tumors
Brief Title: Clinical Trial of Lurbinectedin (PM01183) in Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-B-005-14
Record Dates: First submitted 2015-05-06; First posted 2015-05-27 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — PM 01183

ARMS (1):
- lurbinectedin (PM01183) (Experimental): lurbinectedin (PM01183) 4 mg vials of powder for concentrate for solution for infusion
  Interventions: Drug: lurbinectedin (PM01183)

INTERVENTIONS:
Drug: lurbinectedin (PM01183)

SUMMARY:
Multicenter, open-label, exploratory, phase II clinical trial to evaluate the efficacy and safety of PM01183 in previously treated patients with advanced solid tumors

DETAILED DESCRIPTION:
Patients with relapsed small cell lung cancer (SCLC), head and neck carcinoma (H&N), neuroendocrine tumors (NETs), biliary tract carcinoma, endometrial carcinoma, BRCA 1/2-associated metastatic breast carcinoma, carcinoma of unknown primary site, germ cell tumors (GCTs), and Ewing's family of tumors (EFTs) will be enrolled in nine different cohorts. Up to 25 evaluable patients are planned to be enrolled in each cohort (50 in the endometrial carcinoma and 100 in the SCLC cohort).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Voluntary signed informed consent (IC)
* Pathologically proven diagnosis of any of the following malignancies:

  * Small cell lung cancer (SCLC).
  * Head and neck carcinoma (H&N). Salivary glands tumors are excluded.
  * Neuroendocrine tumors (NETs), grade 2 and grade 3 according to World Health Organization classification.
  * Biliary tract carcinoma.
  * Endometrial carcinoma.
  * BRCA 1/2- associated metastatic breast carcinoma
  * Carcinoma of unknown primary site.
  * Germ cell tumor (GCTs), excluding immature teratoma, or teratoma with malignant transformation.
  * Ewing's family of tumors (EFTs)
* Prior treatment. Patients must have received:

  * SCLC, endometrial carcinoma: one prior chemotherapy-containing line.
  * H&N, NETs, biliary tract, CUP: one or two prior chemotherapy-containing lines
  * GCTs: no limit of prior therapy
  * EFTs: no more than two prior chemotherapy-containing lines in the metastatic/recurrent setting.
  * BRCA 1/2-associated metastatic breast carcinoma: at least one but no more than three prior chemotherapy-containing lines.
* Performance status ≤ 2 [Eastern Cooperative Oncology Group (ECOG)]
* Adequate major organ function
* At least three weeks since the last chemotherapy
* Women of childbearing potential must have pregnancy excluded by appropriate testing before study entry

Exclusion Criteria:

* Prior treatment with PM01183 or trabectedin
* Prior or concurrent malignant disease unless in complete remission for more than five years
* Known central nervous system (CNS) involvement
* Relevant diseases or clinical situations which may increase the patient's risk
* Pregnant or breastfeeding women and fertile patients (men and women) who are not using an effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (7):
  - Sarcoma Oncology Research Center, LLC, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Massachussets General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Centre, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Institute for Drug Development, Cancer Therapy & Research Center at University of Texas Health Science Center, San Antonio, Texas
- Institut Jules Bordet, Brussels, Belgium
- France (3):
  - Hôpital Cochin, Paris
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Charité Universitätsmedizin Berlin - Campus Benjamin Franklin - Comprehensive Cancer Center, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
- Italy (5):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Istituto Ortopedico Rizzoli, Bologna
  - lstituto Europeo di Oncologia, Milan
  - ASST Monza - Ospedale San Gerardo di Monza Struttura Complessa di Oncologia Medica, Monza
  - AUSL Romagna - Ospedale Santa Maria delle Croci, Ravenna
- Spain (18):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hopsital Universitario Donostia - Donostia Unibertsitate Ospitalea, San Sebastián, Guipúzcoa
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario De Navarra, Pamplona, Navarre
  - Hospital Universitario Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall D' Hebron, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Complejo Hospitalario de Especialidades Virgen de la Victoria, Málaga
  - Hospital Universitari i Polotècnic la Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Skane University Hospital, Lund, Sweden
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
- UCL Cancer Institute, London, United Kingdom

REFERENCES:
- [Derived] Kristeleit R, Leary A, Delord JP, Moreno V, Oaknin A, Castellano D, Shappiro GI, Fernandez C, Kahatt C, Alfaro V, Siguero M, Rueda D, Zeaiter A, Awada A, Santaballa A, Zaman K, Sehouli J, Subbiah V. Lurbinectedin in patients with pretreated endometrial cancer: results from a phase 2 basket clinical trial and exploratory translational study. Invest New Drugs. 2023 Oct;41(5):677-687. doi: 10.1007/s10637-023-01383-2. Epub 2023 Aug 9. PMID 37556023
- [Derived] Boni V, Pistilli B, Brana I, Shapiro GI, Trigo J, Moreno V, Castellano D, Fernandez C, Kahatt C, Alfaro V, Siguero M, Zeaiter A, Longo F, Zaman K, Anton A, Paredes A, Huidobro G, Subbiah V. Lurbinectedin, a selective inhibitor of oncogenic transcription, in patients with pretreated germline BRCA1/2 metastatic breast cancer: results from a phase II basket study. ESMO Open. 2022 Oct;7(5):100571. doi: 10.1016/j.esmoop.2022.100571. Epub 2022 Aug 28. PMID 36037567
- [Derived] Longo-Munoz F, Castellano D, Alexandre J, Chawla SP, Fernandez C, Kahatt C, Alfaro V, Siguero M, Zeaiter A, Moreno V, Sanz-Garcia E, Awada A, Santaballa A, Subbiah V. Lurbinectedin in patients with pretreated neuroendocrine tumours: Results from a phase II basket study. Eur J Cancer. 2022 Sep;172:340-348. doi: 10.1016/j.ejca.2022.06.024. Epub 2022 Jul 10. PMID 35830841
- [Derived] Subbiah V, Brana I, Longhi A, Boni V, Delord JP, Awada A, Boudou-Rouquette P, Sarantopoulos J, Shapiro GI, Elias A, Ratan R, Fernandez C, Kahatt C, Cullell-Young M, Siguero M, Zeaiter A, Chawla SP. Antitumor Activity of Lurbinectedin, a Selective Inhibitor of Oncogene Transcription, in Patients with Relapsed Ewing Sarcoma: Results of a Basket Phase II Study. Clin Cancer Res. 2022 Jul 1;28(13):2762-2770. doi: 10.1158/1078-0432.CCR-22-0696. PMID 35486638
- [Derived] Fernandez-Teruel C, Fudio S, Lubomirov R. Integrated exposure-response analysis of efficacy and safety of lurbinectedin to support the dose regimen in small-cell lung cancer. Cancer Chemother Pharmacol. 2022 May;89(5):585-594. doi: 10.1007/s00280-021-04366-3. Epub 2021 Nov 5. PMID 34739582
- [Derived] Subbiah V, Paz-Ares L, Besse B, Moreno V, Peters S, Sala MA, Lopez-Vilarino JA, Fernandez C, Kahatt C, Alfaro V, Siguero M, Zeaiter A, Zaman K, Lopez R, Ponce S, Boni V, Arrondeau J, Delord JP, Martinez M, Wannesson L, Anton A, Valdivia J, Awada A, Kristeleit R, Olmedo ME, Rubio MJ, Sarantopoulos J, Chawla SP, Mosquera-Martinez J, D' Arcangelo M, Santoro A, Villalobos VM, Sands J, Trigo J. Antitumor activity of lurbinectedin in second-line small cell lung cancer patients who are candidates for re-challenge with the first-line treatment. Lung Cancer. 2020 Dec;150:90-96. doi: 10.1016/j.lungcan.2020.10.003. Epub 2020 Oct 10. PMID 33096421
- [Derived] Trigo J, Subbiah V, Besse B, Moreno V, Lopez R, Sala MA, Peters S, Ponce S, Fernandez C, Alfaro V, Gomez J, Kahatt C, Zeaiter A, Zaman K, Boni V, Arrondeau J, Martinez M, Delord JP, Awada A, Kristeleit R, Olmedo ME, Wannesson L, Valdivia J, Rubio MJ, Anton A, Sarantopoulos J, Chawla SP, Mosquera-Martinez J, D'Arcangelo M, Santoro A, Villalobos VM, Sands J, Paz-Ares L. Lurbinectedin as second-line treatment for patients with small-cell lung cancer: a single-arm, open-label, phase 2 basket trial. Lancet Oncol. 2020 May;21(5):645-654. doi: 10.1016/S1470-2045(20)30068-1. Epub 2020 Mar 27. PMID 32224306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient registration was on 25 August 2015 and the first study treatment administration was on 25 August 2015. The last patient registration was on 30 November 2018 and the last study treatment administration was on 29 November 2019. The date of last follow-up (cutoff-date) was 18 September 2020.
Groups:
- Biliary Tract Carcinoma Cohort: Patients with Pathologically proven diagnosis of biliary tract carcinoma
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Carcinoma of Unknown Primary Site Cohort: Patients with pathologically proven diagnosis of carcinoma of unknown primary site
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Endometrial Carcinoma Cohort: Patients with pathologically proven diagnosis of endometrial carcinoma
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Ewing's Family of Tumors Cohort: Patients with pathologically proven diagnosis of Ewing's Family of Tumors
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Germ Cell Tumors Cohort: Patients with pathologically proven diagnosis of Germ Cell Tumors, excluding immature teratoma, or teratoma with malignant transformation.
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Head and Neck Carcinoma Cohort: Patients with Pathologically proven diagnosis of Head and Neck Carcinoma. Salivary glands tumors were excluded.
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- BRCA1/2-associated Metastatic Breast Carcinoma Cohort: Patients with pathologically proven diagnosis of BRCA1/2-associated metastatic breast carcinoma
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Neuroendocrine Tumors Cohort: Patients with Pathologically proven diagnosis of Neuroendocrine Tumors, grade 2 and 3 according to World Health Organization (WHO) classification.
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
- Small Cell Lung Cancer Cohort: Patients with pathologically proven diagnosis of small cell lung cancer
  Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m^2. Dose was capped at body surface area (BSA) of 2.0 m^2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
Period: Overall Study
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Started | 19 | 19 | 76 | 29 | 24 | 15 | 21 | 32 | 110
Treated | 19 | 19 | 73 | 28 | 23 | 15 | 21 | 32 | 105
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 19 | 19 | 76 | 29 | 24 | 15 | 21 | 32 | 110
Not completed — Progressive disease | 17 | 16 | 59 | 23 | 16 | 12 | 19 | 27 | 0
Not completed — Death | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 95
Not completed — Physician Decision | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Non treatment-related adverse event | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Treatment-related adverse events | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 0
Not completed — Patient moves to compassionate use | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 5 | 2 | 3 | 2 | 0 | 1 | 2
Not completed — Multiple delay/holds on treatment | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Never treated | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Study termination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Treated patients only
Groups:
- Biliary Tract Carcinoma Cohort: Patients with Pathologically proven diagnosis of biliary tract carcinoma
- Carcinoma of Unknown Primary Site Cohort: Patients with pathologically proven diagnosis of carcinoma of unknown primary site
- Endometrial Carcinoma Cohort: Patients with pathologically proven diagnosis of endometrial carcinoma
- Ewing's Family of Tumors Cohort: Patients with pathologically proven diagnosis of Ewing's Family of Tumors
- Germ Cell Tumors Cohort: Patients with pathologically proven diagnosis of Germ Cell Tumors, excluding immature teratoma, or teratoma with malignant transformation.
- Head and Neck Carcinoma Cohort: Patients with Pathologically proven diagnosis of Head and Neck Carcinoma. Salivary glands tumors were excluded.
- BRCA1/2-associated Metastatic Breast Carcinoma Cohort: Patients with pathologically proven diagnosis of BRCA1/2-associated metastatic breast carcinoma
- Neuroendocrine Tumors Cohort: Patients with Pathologically proven diagnosis of Neuroendocrine Tumors, grade 2 and 3 according to World Health Organization (WHO) classification.
- Small Cell Lung Cancer Cohort: Patients with pathologically proven diagnosis of small cell lung cancer
- Total: Total of all reporting groups
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort | Total
Number analyzed (Participants) | 19 | 19 | 73 | 28 | 23 | 15 | 21 | 32 | 105 | 335
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 37 | 27 | 20 | 9 | 19 | 19 | 68 | 222
  >=65 years | 6 | 9 | 36 | 1 | 3 | 6 | 2 | 13 | 37 | 113
Age, Continuous [Median (Full Range); unit: years] | 61 [34 to 74] | 61 [27 to 78] | 64 [32 to 80] | 33 [18 to 74] | 36 [21 to 73] | 62 [39 to 81] | 45 [29 to 73] | 63 [23 to 77] | 60 [40 to 83] | 60 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 73 | 12 | 7 | 1 | 21 | 12 | 42 | 189
  Male | 9 | 8 | 0 | 16 | 16 | 14 | 0 | 20 | 63 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 15 | 45 | 21 | 15 | 12 | 18 | 24 | 79 | 242
  Black of African American | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 1 | 7
  Asian | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 6
  American Indian or Alaska native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not race available | 6 | 4 | 22 | 4 | 7 | 2 | 3 | 7 | 24 | 79
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Belgium | 2 | 2 | 3 | 1 | 0 | 0 | 0 | 2 | 3 | 13
  United States | 3 | 6 | 17 | 16 | 12 | 4 | 2 | 6 | 11 | 77
  Italy | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 6
  United Kingdom | 0 | 1 | 9 | 0 | 0 | 0 | 0 | 0 | 3 | 13
  France | 4 | 2 | 17 | 3 | 6 | 2 | 3 | 5 | 20 | 62
  Switzerland | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 7 | 10
  Germany | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Spain | 10 | 8 | 23 | 5 | 4 | 9 | 15 | 18 | 59 | 151
Eastern Cooperative Oncology Group performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 5 | 8 | 32 | 11 | 2 | 5 | 18 | 8 | 38 | 127
    1 | 14 | 10 | 35 | 16 | 19 | 10 | 2 | 23 | 59 | 188
    2 | 0 | 1 | 6 | 1 | 2 | 0 | 1 | 1 | 8 | 20
Weight [Median (Full Range); unit: kg] | 72.2 [45.0 to 115.0] | 65.0 [50.1 to 108.2] | 70.0 [42.5 to 140.8] | 77.0 [51.0 to 127.7] | 78.5 [59.0 to 116.3] | 73.0 [49.0 to 107.0] | 65.5 [52.0 to 115.1] | 64.0 [47.0 to 121.0] | 71.0 [46.0 to 138.3] | 71.0 [42.5 to 140.8]
Height [Median (Full Range); unit: cm] | 168 [148 to 187] | 164.5 [141 to 187] | 161 [143 to 180] | 173 [155 to 193] | 177 [157 to 190] | 170 [155 to 186] | 163.0 [147 to 177] | 169 [150 to 190] | 167 [150 to 183] | 165 [141 to 193]
Body surface area [Median (Full Range); unit: m^2] | 1.9 [1.4 to 2.4] | 1.8 [1.5 to 2.4] | 1.8 [1.3 to 2.6] | 1.9 [1.6 to 2.4] | 2.0 [1.7 to 2.4] | 1.8 [1.5 to 2.2] | 1.7 [1.5 to 2.1] | 1.7 [1.4 to 2.5] | 1.8 [1.4 to 2.6] | 1.8 [1.3 to 2.6]
Albumin [Median (Full Range); unit: g/dL] | 3.7 [2.9 to 4.7] | 3.7 [3.2 to 4.4] | 4.1 [2.7 to 4.7] | 4.2 [3.3 to 4.9] | 4.1 [3.2 to 4.8] | 3.8 [3.0 to 4.4] | 4.1 [3.0 to 5.0] | 4.0 [3.1 to 4.6] | 4.1 [3.1 to 5.1] | 4.0 [2.7 to 5.1]
Albumin [Count of Participants; unit: Participants]
  <3.5 g/dL | 5 | 4 | 9 | 2 | 4 | 3 | 1 | 9 | 13 | 50
  ≥3.5 g/dL | 14 | 15 | 64 | 26 | 19 | 12 | 20 | 23 | 92 | 285
Stage at diagnosis [Count of Participants; unit: Participants]
  Early | 0 | 0 | 23 | 14 | 8 | 4 | 10 | 5 | 3 | 67
  Locally advanced | 4 | 0 | 27 | 5 | 1 | 7 | 6 | 8 | 29 | 87
  Metastatic | 15 | 19 | 23 | 9 | 14 | 4 | 5 | 19 | 73 | 181
Number of sites at baseline [Median (Full Range); unit: sites at baseline] | 3 [2 to 6] | 2 [1 to 4] | 2 [1 to 7] | 2 [1 to 6] | 3 [1 to 4] | 2 [1 to 6] | 2 [1 to 4] | 3 [1 to 7] | 3 [1 to 6] | 3 [1 to 7]
Sites at baseline [Count of Participants; unit: Participants]
  <3 sites | 6 | 12 | 40 | 18 | 7 | 10 | 12 | 13 | 26 | 144
  ≥3 sites | 13 | 7 | 33 | 10 | 16 | 5 | 9 | 19 | 79 | 191
Time from diagnosis to registration [Median (Full Range); unit: months] | 8.4 [3.8 to 23.0] | 10.8 [4.6 to 62.9] | 18.4 [4.3 to 190.9] | 28.6 [6.9 to 140.5] | 48.2 [7.3 to 308.8] | 19.5 [2.9 to 426.1] | 50.1 [16.2 to 236.0] | 13.3 [3.0 to 93.2] | 8.2 [2.1 to 20.0] | 13.7 [2.1 to 426.1]
Time from advanced disease to registration [Median (Full Range); unit: month] | 10.6 [6.3 to 23.0] | NA [NA to NA] — All patients were metastatic | 17.5 [0.9 to 97.0] | 20.4 [0.4 to 54.2] | 33.5 [10.7 to 86.8] | 18.4 [9.7 to 72.7] | 31.9 [14.1 to 115.9] | 17.2 [3.8 to 93.2] | 9.1 [0.3 to 20.0] | 15.0 [0.3 to 115.9]
Prior surgery [Count of Participants; unit: Participants] | 2 | 2 | 62 | 20 | 21 | 9 | 19 | 11 | 2 | 148
Prior radiotherapy [Count of Participants; unit: Participants] | 2 | 8 | 39 | 20 | 7 | 11 | 20 | 7 | 76 | 190
Systemic lines [Count of Participants; unit: Participants]
  1 line | 13 | 12 | 54 | 5 | 0 | 5 | 0 | 14 | 98 | 201
  2 lines | 6 | 7 | 15 | 15 | 4 | 8 | 7 | 13 | 7 | 82
  3 lines | 0 | 0 | 3 | 5 | 8 | 2 | 7 | 4 | 0 | 29
  4 or more lines | 0 | 0 | 1 | 3 | 11 | 0 | 7 | 1 | 0 | 23
Advanced chemotherapy lines [Count of Participants; unit: Participants]
  0 lines | 19 | 0 | 15 | 5 | 0 | 0 | 1 | 0 | 105 | 145
  1 line | 0 | 12 | 47 | 7 | 1 | 5 | 5 | 17 | 0 | 94
  2 lines | 0 | 7 | 8 | 13 | 4 | 9 | 7 | 10 | 0 | 58
  3 lines | 0 | 0 | 2 | 3 | 8 | 1 | 6 | 4 | 0 | 24
  4 or more lines | 0 | 0 | 1 | 0 | 10 | 0 | 2 | 1 | 0 | 14
Best response to last therapy [Count of Participants; unit: Participants] — According to the RECIST v.1.1, Complete Response: Disappearance of all target lesions; Partial Response (PR): ≥30% decrease in the sum of the longest diameters of target lesions compared with baseline; Progressive disease (PD): ≥20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest; diameter recorded or the appearance of one or more new lesions; Stable Disease: Neither PR or PD
  Participants
    Complete response | 0 | 3 | 7 | 0 | 0 | 0 | 1 | 0 | 9 | 20
    Partial reponse | 4 | 4 | 20 | 0 | 2 | 5 | 2 | 5 | 70 | 112
    Stable disease | 7 | 5 | 13 | 0 | 5 | 2 | 6 | 14 | 19 | 71
    Progression disease | 8 | 4 | 15 | 0 | 15 | 7 | 7 | 11 | 4 | 71
    Unknown | 0 | 3 | 18 | 28 | 1 | 1 | 5 | 2 | 3 | 61
Time to progression to last prior therapy [Median (Full Range); unit: months] | 5.2 [1.0 to 14.0] | 3.9 [0.9 to 22.9] | 8.0 [1.4 to 23.5] | 8.7 [0.4 to 25.8] | 2.7 [0.8 to 29.6] | 4.6 [1.4 to 26.1] | 5.0 [1.3 to 32.1] | 3.6 [1.1 to 24.0] | 6.5 [1.4 to 17.8] | 6.4 [0.4 to 32.1]
Time from last progression disease before study entry [Median (Full Range); unit: weeks] | 3.0 [0.3 to 6.7] | 2.6 [0.1 to 33.7] | 2.9 [0.0 to 24.6] | 2.1 [0.0 to 7.1] | 1.4 [0.3 to 6.4] | 2.4 [0.0 to 24.7] | 1.6 [0.1 to 7.6] | 2.6 [0.6 to 21.9] | 1.6 [0.0 to 10.0] | 2.1 [0.0 to 33.7]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate was defined as the percentage of patients with a confirmed response, either CR or PR, according to the RECIST v.1.1. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥30% decrease in the sum of the longest diameters of target lesions compared with baseline; Progressive disease: ≥20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest; diameter recorded or the appearance of one or more new lesions; Stable Disease: Neither PR or PD
Time Frame: From the start of treatment to the date of progression or the start of a subsequent therapy or end of patient's follow-up, until Cycle 6 (21-day cycle)
Population: Treated patients and with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of participants | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 17.6] | 11.3 [5.0 to 21.0] | 14.3 [4.0 to 32.7] | 4.3 [0.1 to 21.9] | 0.0 [0.0 to 24.7] | 28.6 [11.3 to 55.2] | 6.5 [0.8 to 21.4] | 36.2 [27.0 to 46.1]

2. Primary Outcome: Response by Investigator Assessment
Description: When response is the primary endpoint, and thus all patients must have measurable disease to enter the trial, all patients included in the study must be accounted for in the report of the results, even if there are major protocol treatment deviations or if they are not evaluable. Each patient will be assigned one of the following: Complete Response: Disappearance of all target lesions; Partial Response: ≥30% decrease in the sum of the longest diameters of target lesions; Progressive disease: ≥20% increase in the sum of the longest diameter of target lesions; diameter recorded or the appearance of one or more new lesions; Stable Disease: Neither PR or PD; Inevaluable for response: specify reasons (for example: early death, malignant disease, toxicity; tumour assessments not repeated/incomplete; other).
  Normally, all eligible patients should be included in the denominator for the calculation of the response rate for phase II trials.
Time Frame: as for outcome 1
Population: Treated patients with disease measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
Participants
  Complete Response | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 6 | 4 | 1 | 0 | 6 | 2 | 38
  Stable Disease | 5 | 11 | 29 | 12 | 8 | 3 | 10 | 9 | 34
  Progressive disease | 11 | 7 | 30 | 9 | 12 | 8 | 5 | 18 | 28
  Inevaluable for response | 1 | 1 | 4 | 3 | 2 | 2 | 0 | 2 | 5

3. Secondary Outcome: Duration of Response
Description: Duration of Response by Investigator's Assessment, defined as the time between the date when the response criteria (PR or CR, whichever one is first reached) are fulfilled to the first date when disease progression (PD), recurrence or death is documented.
Time Frame: as for outcome 1
Population: Patients with response to treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 1 | 0 | 8 | 4 | 1 | 0 | 6 | 2 | 38
months | 3.4 [NA to NA] — Only 1 patient |  | 9.2 [3.4 to 18.0] | 4.2 [2.9 to 5.5] | 10.6 [NA to NA] — Only 1 patient |  | 8.6 [2.9 to NA] — Not reached | 4.7 [4.0 to 5.4] | 5.3 [4.1 to 6.2]

4. Secondary Outcome: Clinical Benefit
Description: Clinical Benefit Rate was defined as Overall Response Rate or Stable Disease lasting over four months (SD ≥ 4 months)
Time Frame: as for outcome 1
Population: Treated patients with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of participants | 11.1 [1.4 to 34.7] | 36.8 [16.3 to 61.6] | 35.2 [24.2 to 47.5] | 39.3 [21.5 to 59.4] | 26.1 [10.2 to 48.4] | 15.4 [1.9 to 45.4] | 57.1 [34.0 to 78.2] | 29.0 [14.2 to 48.0] | 45.7 [36.0 to 55.7]

5. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate was defined as Overall Response Rate or Stable Disease
Time Frame: From the start of treatment to the date of progression or the start of a subsequent therapy or end of patient's follow-up, until Cycle 6
Population: Treated patients with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of paticipants | 33.3 [13.3 to 59.0] | 57.9 [33.5 to 79.7] | 52.1 [39.9 to 64.1] | 57.1 [37.2 to 75.5] | 39.1 [19.7 to 61.5] | 23.1 [5.0 to 53.8] | 76.2 [52.8 to 91.8] | 35.5 [19.2 to 54.6] | 68.6 [58.8 to 77.3]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free Survival (PFS), defined as the period of time from the date of first infusion to the date of PD, death (of any cause), or last tumor evaluation.
  Progressive disease: ≥20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest
Time Frame: From the date of first infusion to the date of progression disease, death (of any cause), or last tumor evaluation, up to an average of 5 years
Population: Treated patients with disease measurement
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
months | 1.3 [1.1 to 2.5] | 2.7 [1.3 to 4.4] | 2.6 [1.4 to 4.0] | 2.7 [1.4 to 4.3] | 1.5 [0.9 to 8.9] | 1.3 [1.2 to 2.1] | 4.1 [2.3 to 6.5] | 1.4 [1.2 to 3.0] | 3.7 [2.6 to 4.3]

7. Secondary Outcome: Progression-free Survival at 4 Months
Description: Progression-free Survival at 4, defined as the probability of being free from progression and death after the first infusion at 4 months. Progressive disease: ≥20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest
Time Frame: At 4 months
Population: Treated patients with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of participants | 13.7 [0.0 to 31.1] | 38.9 [16.4 to 61.4] | 39.7 [28.2 to 51.3] | 46.2 [27.0 to 65.3] | 30.7 [11.0 to 50.4] | 15.4 [0.0 to 35.0] | 57.1 [36.0 to 78.3] | 30.0 [13.6 to 46.4] | 46.5 [36.8 to 56.3]

8. Secondary Outcome: Progression-free Survival at 6 Months
Description: Progression-free Survival at 6, defined as the probability of being free from progression and death after the first infusion at 6 months. Progressive disease: ≥20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest
Time Frame: At 6 months
Population: Treated patients with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of participants | 13.7 [0.0 to 31.1] | 22.2 [3.0 to 41.4] | 29.0 [18.2 to 39.8] | 23.1 [5.9 to 40.3] | 30.7 [11.0 to 50.4] | 7.7 [0.0 to 22.2] | 33.3 [13.2 to 53.5] | 16.7 [3.3 to 30.0] | 33.4 [24.1 to 42.6]

9. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the period of time from the date of first infusion to the date of death or last contact in case of patients lost to follow-up or alive at the clinical cutoff established for the cohort.
Time Frame: From the date of first infusion to the date of death or last contact, up to an average of 5 years
Population: Treated patients with disease measurement
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
months | 7.3 [2.7 to 8.9] | 7.7 [3.8 to 18.8] | 9.3 [6.1 to 12.8] | 12.0 [8.5 to 18.5] | 9.2 [2.7 to 17.4] | 5.7 [2.1 to 12.1] | 16.1 [8.7 to NA] — Not reached | 7.4 [3.4 to 16.2] | 8.1 [6.5 to 10.9]

10. Secondary Outcome: Overall Survival at 6 Months
Description: Overall Survival at 6 months defined as the probability of being alive after the first infusion at 6 months
Time Frame: At 6 months
Population: Treated patients with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of participants | 58.2 [34.5 to 82.0] | 55.6 [32.6 to 78.5] | 62.8 [51.2 to 74.4] | 88.2 [75.7 to 100.0] | 55.0 [32.8 to 77.1] | 38.5 [12.0 to 64.9] | 79.2 [61.0 to 97.4] | 52.1 [33.9 to 70.3] | 68.6 [59.5 to 77.6]

11. Secondary Outcome: Overall Survival at 12 Months
Description: Overall Survival at 12 months defined as the probability of being alive after the first infusion at 12 months
Time Frame: At 12 months
Population: Treated patients with disease measurement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Biliary Tract Carcinoma Cohort | Carcinoma of Unknown Primary Site Cohort | Endometrial Carcinoma Cohort | Ewing's Family of Tumors Cohort | Germ Cell Tumors Cohort | Head and Neck Carcinoma Cohort | BRCA1/2-associated Metastatic Breast Carcinoma Cohort | Neuroendocrine Tumors Cohort | Small Cell Lung Cancer Cohort
Number analyzed (Participants) | 18 | 19 | 71 | 28 | 23 | 13 | 21 | 31 | 105
percentage of participants | 21.8 [0.4 to 43.3] | 36.5 [13.1 to 59.8] | 45.8 [33.8 to 75.9] | 48.5 [27.8 to 69.2] | 34.4 [11.3 to 57.4] | 30.8 [5.7 to 55.9] | 58.1 [35.9 to 80.2] | 38.2 [20.5 to 55.9] | 34.8 [25.5 to 44.1]

ADVERSE EVENTS:
Time Frame: From the date of first infusion to the date of death or last contact, up to an average of 5 years
Description: Safety in the entire trial population is a secondary objective defined in the protocol as all patients were exposed to the same unique dose of lurbinectedin. Consequently, adverse events are reported in a combined mode for all groups (cohorts) to provide a clear picture of the drug safety in the whole population.
  Out of the 345 patients enrolled there were 10 patients who did not receive lurbinectedin treatment so patients at risk is 335 (345-10)
Groups:
- Lurbinectedin (PM01183): Lurbinectedin was administered over a minimum total volume of 100 mL of solution for infusion (either on 5% glucose or 0.9% sodium chloride), through a central catheter, or over a minimum total volume of 250 mL if administered through a peripheral line, always over one hour at a fixed infusion rate. Starting dose was 3.2 mg/m2. Dose was capped at body surface area (BSA) of 2.0 m2 (i.e., dose did not exceed 6.4 mg).
  Patients received lurbinectedin intravenously (i.v.) as a one-hour infusion on Day 1 q3wk (three weeks = one treatment cycle).
Arm/Group | Lurbinectedin (PM01183)
All-Cause Mortality (participants affected / at risk) | 261/335
Serious Adverse Events (participants affected / at risk) | 136/335
Other Adverse Events (participants affected / at risk) | 330/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurbinectedin (PM01183) (N=335)
Anaemia (Blood and lymphatic system disorders) | 10 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 (21)
Leukopenia (Blood and lymphatic system disorders) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 15 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (36)
Tachycardia (Cardiac disorders) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (12)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 4 (5)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 7 (9)
Asthenia (General disorders) | 2 (2)
Gait disturbance (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 15 (21)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 6 (8)
Cholangitis (Hepatobiliary disorders) | 3 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (10)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood phosphorus decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Aphasia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hemiplegia (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2)
Subacute combined cord degeneration (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (5)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cementoplasty (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 2 (2)
Superior vena cava occlusion (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurbinectedin (PM01183) (N=335)
Anaemia (Blood and lymphatic system disorders) | 59 (100)
Neutropenia (Blood and lymphatic system disorders) | 89 (174)
Abdominal pain (Gastrointestinal disorders) | 54 (83)
Abdominal pain upper (Gastrointestinal disorders) | 19 (21)
Constipation (Gastrointestinal disorders) | 116 (189)
Diarrhoea (Gastrointestinal disorders) | 62 (104)
Nausea (Gastrointestinal disorders) | 167 (276)
Vomiting (Gastrointestinal disorders) | 76 (126)
Asthenia (General disorders) | 129 (335)
Chest pain (General disorders) | 23 (28)
Fatigue (General disorders) | 122 (242)
Mucosal inflammation (General disorders) | 19 (23)
Oedema peripheral (General disorders) | 30 (35)
Pyrexia (General disorders) | 48 (56)
Weight decreased (Investigations) | 25 (33)
Decreased appetite (Metabolism and nutrition disorders) | 102 (144)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 51 (71)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (32)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (34)
Headache (Nervous system disorders) | 25 (28)
Neuropathy peripheral (Nervous system disorders) | 19 (27)
Insomnia (Psychiatric disorders) | 34 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 58 (71)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 77 (99)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02454972/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT02454972/SAP_001.pdf